CLINICAL TRIAL: NCT04151446
Title: Evaluation of the Safety & Efficacy of the Laser Scleral Microporation Procedure to Restore Visual Function and Range of Accommodation
Brief Title: Safety & Efficacy of the Laser Scleral Microporation Procedure (Taiwan)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate Enrollment
Sponsor: ACE Vision Group, Inc. (Industry)
Collaborators: Vision Renu Taiwan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TWAVG-2017-01
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2021-10

CONDITIONS: Presbyopia
Keywords: Presbyopia; Sclera; Laser Scleral Microporation
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser Scleral Microporation procedure (Experimental): Patients suffering from presbyopia will receive bilateral Laser Scleral Microporation procedure.
  Interventions: Device: Laser Scleral Microporation

INTERVENTIONS:
Device: Laser Scleral Microporation — Partial depth scleral microporations with an Er:YAG laser in a predetermined pattern.

SUMMARY:
A new minimally invasive procedure for treating presbyopia is being evaluated to determine if there is improvement in near and intermediate vision after treatment.

DETAILED DESCRIPTION:
This is a prospective, controlled, single-center clinical study to evaluate the safety and efficacy of the Laser Scleral Microporation Procedure.

Laser Scleral Microporation Procedure is a treatment to restore visual and accommodative function in presbyopic patients. The subjects are bilaterally treated with the Laser Scleral Microporation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand and sign an informed consent;
2. Willing and able to attend postoperative examinations per protocol schedule;
3. 45 years of age or greater, of either gender or any race;
4. Less than (<) 1.00D of astigmatism in each eye, measured in their manifest refraction;
5. Mean refractive spherical equivalent refraction (MRSE) of +/- 0.50D for distance vision; Note: Subjects who meet this criterion as a result of prior laser refractive surgery (LASIK, LASEK or PRK) may qualify; however, the subject must have had the LVC procedure performed at least 12 months prior to the Laser Scleral Microporation procedure and be stable.
6. Uncorrected distance visual acuity (UDVA) is better than or equal to 20/40 (logMAR 0.30) in each eye, and a Corrected Distance Visual Acuity (CDVA) is better than or equal to 20/25 (logMAR 0.10) in each eye;
7. Demonstrate Stereopsis of 100 seconds of arc or better using a Randot stereoscopic fly test and reading correction;
8. In good ocular health with the exception of presbyopia;
9. Presbyopia as demonstrated by:

   1. Currently wearing reading glasses and/or bifocals with an ADD of +1.50D or more at 40 cm in each eye; and
   2. Reduced near visual acuity at 40 cm when corrected for distance (DCNVA) of 20/50 (logMAR 0.40) or worse in each eye;
10. Intraocular pressure (IOP) >11mmHg and < 30 mmHg in each eye without IOP-lowering medication;
11. Less than or equal to (≤) 0.50D difference between the manifest refraction and the cycloplegic refraction;
12. Stable distance refraction is present, defined as ≤ 0.50D variation of refraction in the 12 months prior to the Laser Scleral Microporation procedure. Manifest refraction cannot vary more than 0.50D from current spectacles that are at least 12 months of age, or from a documented refraction at least 12 months prior to the preoperative baseline exam; if baseline data is available.
13. Completed a washout period of two weeks (14 days) prior to Laser Scleral Microporation procedure from prior treatment with:

    * With prior medical clearance: NSAIDS, blood thinners, aspirin, and other substances which may increase bleeding;
    * Anti-oxidants, which could affect blood thinning14

      * Any anti-oxidant supplements (e.g., Vitamin B6, Vitamin B12, Vitamin E, Vitamin C, Acai, Ocuvite, etc);
      * Anti-oxidant food supplements, such as shitake mushroom, mushroom extract and oral anti-oxidants.

Exclusion Criteria:

1. Self-reported current pregnancy or breast-feeding, or plans to become pregnant during the entire study period;
2. History of ocular trauma or prior ocular surgery, or expected to require retinal laser treatment or other ocular surgical intervention;
3. Presence of ocular pathology other than cataract such as:

   * Amblyopia or strabismus
   * Corneal abnormalities or disease
   * Dry Eye, presenting with corneal staining15
   * Pupil abnormalities (e.g., corectopia, Adie's)
   * Capsule or zonular abnormalities
   * Intraocular inflammation
   * Retinal disease or pathology
   * Glaucoma (any type)
   * History of prior ocular surgery other than keratorefractive surgery;
4. Known pathology that may affect visual acuity and/or are predicted to cause future acuity losses to a level of 20/30 (logMAR 0.18) or worse (e.g., macular degeneration);
5. Previous corneal surgery (e.g., corneal transplant, DSAEK/DSEK, lamellar keratoplasty), except for LASIK, EpiLASIK/LASEK, or PRK;
6. Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy);
7. Keratoconus or keratoconus suspect with CDVA of less than (<) 20/20 (< logMAR 0.00) at distance;
8. Near visual acuity at 40cm equivalent to their distance vision with distance correction (i.e., no evident effect of reduced accommodative range);
9. Use of systemic or ocular medications that may affect vision (the use of any miotic or cycloplegic agent is specifically contraindicated);
10. Acute or chronic disease or illness that could increase the operative risk or confound the study outcome(s) (e.g., diabetes mellitus, immunocompromised, connective tissue disease);
11. Uncontrolled systemic or ocular disease;
12. Any abnormality preventing reliable applanation tonometry in EITHER eye;
13. Undilatable pupil such that one cannot examine the periphery of the retina;
14. Functional eye preference, defined as phoria measuring over 15dp horizontally and/or over 2dp vertically, any strabismus, or suppression.
15. History of scleral ectasia, scleritis, or episcleritis
16. History of nuclear sclerosis LOCS III grade 2 or worse and/or other cataracts reducing CDVA;
17. Known allergies to study medications including topical steroids, antibiotics and NSAIDS;
18. Too thin sclera thickness
19. Per PI discretion, as described below:

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Binocular Uncorrected Near Visual Acuity (UNVA) @ 40cm | 12 months postoperative
  Binocular UNVA is measured with ETDRS charts placed in 40cm distance. This assessment is performed under photopic lighting conditions.

SECONDARY OUTCOMES:
Patient Self-Reporting Questionnaire 1 | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  Outcomes measures of a questionnaire to address the general patient satisfaction and possible side effects of the treatment. For this study, the validated and verified Near Activity Visual Questionnaire (NAVQ) will be used [see citation 1, Buckhurst et al.].
  This questionnaire consists of 10 questions. Each question can be answered with scores between 0 (best outcome and 3 (worst outcome). The answers will be converted to Rasch score according to the NAVQ guidelines.
Patient Self-Reporting Questionnaire 2 | 3 Day, 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  A self-reporting questionnaire will be used to assess adverse events and side effects.
Monocular & Binocular Uncorrected Distance Visual Acuity (UDVA) @ 4m | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance. This assessment is performed monocularly, then binocularly under photopic lighting conditions.
Monocular & Binocular Uncorrected Intermediate Visual Acuity (UIVA) @ 60cm | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  UIVA is measured with ETDRS charts placed in 60cm distance. This assessment is performed monocularly, then binocularly under photopic lighting conditions.
Monocular & Binocular Uncorrected Near Visual Acuity (UNVA) @ 40cm | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  UNVA is measured with ETDRS charts placed in 40cm distance. This assessment is performed monocularly, then binocularly under photopic lighting conditions.
Manifest Refraction | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  This is the manual way to determine the best lenses, by placing carious lenses in front of the subject's eyes and asking questions by using a phoropter. Perform maximum plus subjective refraction with 100% contrast ETDRS cart at 4m. The data contains value for sphere, cylinder and axis cylinder. This assessment is performed under photopic lighting conditions
Monocular & Binocular Best Corrected Distance Visual Acuity (CDVA) @ 4m | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance using best aided corrective glasses. This assessment is performed monocularly, then binocularly under photopic lighting conditions.
Monocular & Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) @ 60cm | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  DCIVA is measured with ETDRS charts placed in 60cm distance using corrective glasses for far distance. This assessment is performed monocularly, then binocularly under photopic lighting conditions.
Monocular & Binocular Distance Corrected Near Visual Acuity (DCNVA) @ 40cm | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  DCNVA is measured with ETDRS charts placed in 40cm distance using corrective glasses for far distance. This assessment is performed monocularly, then binocularly under photopic lighting conditions.
Determination of reading prescription | 1 week; 1 month; 3 months; 6 months ; 12 months; 18 months & 24 months postoperative
  Subjects will be refracted at 40cm based upon distance prescription. The subject holds a near card (Chart 1) at 40cm. With the subject's binocular distance refraction in place, plus power is increased in +0.25 increments binocularly until the subject can read the 0.0 logMAR line on the chart. If the subject cannot read the logMAR 0.0 line with a +2.5D ADD, +2.5D ADD with the visual acuity will be recorded. This assessment will be performed under photopic lighting conditions.
Accommodative Amplitude using binocular & monocular minus lens to blur | 1 week; 1 month; 3 months; 6 months; 12 months & 24 months postoperative
  The amplitude of accommodation will be assessed at distance with introduction of minus power over the distance prescription to stimulate accommodation. The subject will be instructed to focus on the distance Hart chart and slowly add minus power in -0.25D steps until the subject reports first sustained blur on the line. Record the dioptric value where the subject reports the first sustained blur. Subtract the distance prescription from this value to obtain the accommodative amplitude using this method. This test is repeated three times. This assessment is performed binocularly, then monocularly under photopic lighting conditions.
iReST reading test | 1 week; 1 month; 3 months; 6 months; 12 months & 24 months postoperative
  The reading speed will be measured using the International Reading Speed Texts (iReST™), a standardized assessment of reading speed. For this test, the reading prescription determined at each visit will be used and the assessment will be performed under photopic lighting conditions.
Wavefront Aberrometry | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  The iTrace (Tracey Technologies, Houston, TX) measures aberrometry at distance, 60cm and 40cm. Measurements will be performed uncorrected and corrected aided using the distance prescription based upon the manifest refraction. Coma, Spherical Aberration, and Trefoil exams will also be recorded at distance, 60cm and 40cm.
Auto-Keratometry | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  An auto keratometer uses a microprocessor computer to facilitate the rapid measurement of the corneal curvature. The simulated keratometry (Sim K) us determined as the average keratometry, calculated by using the standard keratometric index and the radius of anterior corneal curvature using the the iTrace (Tracey Technologies, Houston TX).
Corneal Topography | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  Corneal topography is a computer assisted diagnostic tool that creates a three-dimensional map of the surface curvature of the cornea. Anterior surface corneal topography using placido disc will be measured using the iTrace unit (Tracey Technologies, Houston, TX).
Speedy-i Accommodation Testing | 1 week; 1 month; 3 months; 6 months; 12 months & 24 months postoperative
  Speedy-i is used for accommodation test and subject's individual Accommodative Micro Fluctuation (AMF) is analyzed.
Stereoacuity | 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  Stereoacuity will be measured under photopic conditions using a standard randot stereoscopic test at 40cm with the subject's reading prescription (determined at each visit). This assessment will be performed under photopic lighting conditions.
Pupillometry | 1 day, 3 day, 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  Measurement of pupil size will be performed under photopic and mesopic lighting conditions. The Neuroptics VIP® -200 pupillometer or equivalent is being used.
Contrast Sensitivity | 1 month; 12 months & 24 months postoperative
  Contrast sensitivity is the subject's ability to distinguish the foreground from the background. This will be measured using ETDRS (Precision Vision Chart 2153) optotypes (5 per acuity level) with 10% contrast placed in 4m distance. Distance prescription should be worn. This assessment will be performed monocularly, then binocularly under photopic lighting conditions.
Axial Length Measurement | 1 month; 12 months & 24 months postoperative
  The length of the globe, or "axial length" will be measured using a non-contact optical low-coherence reflectometry. Recommended devices LENSTAR LS900, Alcom) or (IOLMaster version 7.5 or higher, Carl Zeiss Humphrey).
Slit Lamp Examination | 1 day, 3 days, 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  The slit lamp examination is one examination to analyse the integrity of the eye structures.
  With the slit lamp the ophthalmologist can observe the eyes stereoscopically. A focused slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slit lamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slit lamp:
  * Corneal clarity
  * anterior chamber cells
  * anterior chamber flare
  * lens grading using the LOCS III score card
  * Conjunctival/scleral vessel injection
  * Degree of choroidal hue
  * Conjunctival edema
  * Conjunctival hemorrhages
  * Other corneal/conjunctival/scleral observations
  * Dry Eye
  * Other anterior chamber observations
  * Eyelid edema
Intraocular Pressure Measurement | 1 day, 3 days, 1 week; 1 month; 3 months; 6 months; 12 months; 18 months & 24 months postoperative
  Intraocular Pressure will be measured using Goldmann applanation tonometry. Two measurements will be performed per eye at each visit. If there is more than 2mmHg between the two reading, a third reading will be performed. The value will be an average.
Cycloplegic refraction | 1 month; 12 months & 24 months postoperative
  A cycloplegic refraction at distance using 1% cyclopentolate will be performed to determine the absolute refractive error.
Dilated Fundus exam | 1 month; 12 months & 24 months postoperative
  A Dilated Fundus Exam will also be performed to examine the vitreous, optic nerve, blood vessels, macula and retina to identify eye related diseases or anatomical anomalies.

CONTACTS AND LOCATIONS:
Overall Officials: David Ma, MD, Principal Investigator — Chang Gung Memorial Hospital; Arvin Sun, MD, Principal Investigator — Chang Gung Memorial Hospital, Keelung
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Keelung, Keelung
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

REFERENCES:
- [Background] Buckhurst PJ, Wolffsohn JS, Gupta N, Naroo SA, Davies LN, Shah S. Development of a questionnaire to assess the relative subjective benefits of presbyopia correction. J Cataract Refract Surg. 2012 Jan;38(1):74-9. doi: 10.1016/j.jcrs.2011.07.032. Epub 2011 Nov 10. PMID 22078121